CLINICAL TRIAL: NCT00127114
Title: Amantadine for the Treatment of Behavioral Disturbance in Frontotemporal Dementia (FTD)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No funding and exclusion criteria were to stringent.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04033101
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Dementia
Keywords: Behavioral disturbance; Frontotemporal dementia; Dementia; Amantadine; Behavioral disturbance due to frontotemporal dementia
MeSH Terms: conditions — Dementia; Mental Disorders; Frontotemporal Dementia | interventions — Amantadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Amantadine (Experimental)
  Interventions: Drug: Amantadine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amantadine
  Arms: Amantadine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to test whether or not the medication amantadine is effective in reducing behavioral disturbances in patients with frontotemporal dementia.

DETAILED DESCRIPTION:
Behavioral disturbances are a major cause of morbidity in frontotemporal dementia (FTD), yet little is known about the effectiveness of medications to treat these disturbances. Preliminary data suggests that the dopaminergic agent amantadine may reduce these disturbances. This 6-week, prospective, randomized, placebo-controlled trial will compare amantadine to placebo to assess its effectiveness in reducing behavioral symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Frontotemporal dementia meeting diagnostic criteria of the Report of the Work Group on Frontotemporal Dementia and Pick's Disease (McKhann et al, 2001). Diagnosis will be established by clinical interview by a geriatric psychiatrist or neuropsychiatrist, experienced with the diagnosis of FTD. Patients with the language presentation of FTD will be enrolled if their behavioral disturbance meets the inclusion criteria. Use of these diagnostic criteria would allow for enrollment of patients who in a clinical setting carry the diagnosis of: semantic dementia, primary progressive aphasia, cortical-basal degeneration, progressive supranuclear palsy, (amyotrophic lateral sclerosis (ALS) with dementia, and Pick's disease, as all of these diagnoses are now classified under the rubric of FTD.
* Frontal Behavioral Inventory (FBI) disinhibition subscale score of >16 (Kertesz et al,1997; Kertesz et al 2000). Explanation of this subscale is found under outcome measures.
* Men, women and minority groups will be included, ages 40-90 years old.
* Judged by the attending psychiatrist to be in sufficiently good health so as to be treated using the study protocol in usual outpatient care circumstances.
* Patient, caregivers and or legal representatives provide informed consent for participation in the study, using standard Johns Hopkins Division of Geriatric Psychiatry and Neuropsychiatry procedures.
* Caregiver is available who spends at least 10 hours per week with the patient and is able and willing to accompany the patient in the course of the study and to provide collateral information.

Exclusion Criteria:

* Presence of a brain disease that might otherwise fully explain the presence of dementia or behavior disturbance, such as stroke, Parkinson's disease, traumatic brain injury, multiple sclerosis, and the like.
* Treatment with amantadine is contraindicated in the opinion of the study attending psychiatrist. Examples of this would be patients with advanced heart, liver or kidney disease or a seizure disorder. Creatinine clearance >50mL/min will be required, calculated using the Cockcroft-Gault equation.
* Failure of treatment with amantadine for behavior disturbance of FTD in the past.
* Treatment with a medication that would prohibit the safe concurrent use of amantadine.
* Ongoing regular alcohol use and an unwillingness to stop drinking alcohol during the study period.
* Pregnancy or lactation.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2007-07-26 (Actual); Study Completion 2007-07-26 (Actual)

PRIMARY OUTCOMES:
Frontal Behavioral Inventory, disinhibition subscale | 6 weeks

SECONDARY OUTCOMES:
Frontal Behavior Inventory, total score | 6 weeks
Neuropsychiatric Inventory | 6 weeks
Apathy Evaluation Scale | 6 weeks
Cognitive measures - Mini Mental State Exam (MMSE), Trails Making Test A&B (Trails A&B), Verbal fluency, and Stroop test | 6 weeks
Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) measures | 6 weeks
Zarit Burden Interview | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David M Blass, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Outpatient General Clinical Research Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Drayton SJ, Davies K, Steinberg M, Leroi I, Rosenblatt A, Lyketsos CG. Amantadine for executive dysfunction syndrome in patients with dementia. Psychosomatics. 2004 May-Jun;45(3):205-9. doi: 10.1176/appi.psy.45.3.205. PMID 15123844
- [Background] O'Suilleabhain P, Dewey RB Jr. A randomized trial of amantadine in Huntington disease. Arch Neurol. 2003 Jul;60(7):996-8. doi: 10.1001/archneur.60.7.996. PMID 12873857
- [Background] Verhagen Metman L, Morris MJ, Farmer C, Gillespie M, Mosby K, Wuu J, Chase TN. Huntington's disease: a randomized, controlled trial using the NMDA-antagonist amantadine. Neurology. 2002 Sep 10;59(5):694-9. doi: 10.1212/wnl.59.5.694. PMID 12221159
- [Background] Van Reekum R, Bayley M, Garner S, Burke IM, Fawcett S, Hart A, Thompson W. N of 1 study: amantadine for the amotivational syndrome in a patient with traumatic brain injury. Brain Inj. 1995 Jan;9(1):49-53. doi: 10.3109/02699059509004571. PMID 7874096
- [Background] Imamura T, Takanashi M, Hattori N, Fujimori M, Yamashita H, Ishii K, Yamadori A. Bromocriptine treatment for perseveration in demented patients. Alzheimer Dis Assoc Disord. 1998 Jun;12(2):109-13. doi: 10.1097/00002093-199806000-00009. PMID 9651140
- [Background] Kertesz A, Davidson W, McCabe P, Munoz D. Behavioral quantitation is more sensitive than cognitive testing in frontotemporal dementia. Alzheimer Dis Assoc Disord. 2003 Oct-Dec;17(4):223-9. doi: 10.1097/00002093-200310000-00005. PMID 14657786
- [Background] McDowell S, Whyte J, D'Esposito M. Differential effect of a dopaminergic agonist on prefrontal function in traumatic brain injury patients. Brain. 1998 Jun;121 ( Pt 6):1155-64. doi: 10.1093/brain/121.6.1155. PMID 9648550
- [Background] Sjogren M, Minthon L, Passant U, Blennow K, Wallin A. Decreased monoamine metabolites in frontotemporal dementia and Alzheimer's disease. Neurobiol Aging. 1998 Sep-Oct;19(5):379-84. doi: 10.1016/s0197-4580(98)00086-4. PMID 9880039